CLINICAL TRIAL: NCT00568256
Title: Mind/Body Medicine and IBD Flare-Up
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ali Keshavarzian, Dr. Ali Keshavarzian, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07092603; NCT00571532 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; IBD Flare-Up; Stress
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Mind/Body Course
  Interventions: Behavioral: Mind/Body Courses
- Other (Other): Mind/Body Course
  Interventions: Behavioral: Mind/Body Courses

INTERVENTIONS:
Behavioral: Mind/Body Courses — 8-week Mind/Body course held once a week for 2 hours at a time.

SUMMARY:
Ulcerative Colitis is an Inflammatory Bowel disease that is a life-long, relapsing disabling disorder. Current treatments for Ulcerative Colitis are not satisfactory. Most medications provide only partial relief, are not successful for at least 30% of patients, and have major negative side effects. Mounting evidence indicates that stress is one of the important triggers that activates symptoms of ulcerative colitis and therefore causes flare-up. The primary aim of this study is to see if either of two 8-week Mind-Body courses has an effect in reducing stress and affecting the course and severity of UC.

Hypotheses: Stress causes Ulcerative Colitis flare-up and stress reduction will prevent Ulcerative Colitis flare-up.

DETAILED DESCRIPTION:
Methods: We will enroll 100 subjects in a Phase I/IIa randomized, double-blind, placebo-controlled trial. Subjects will be assigned to one of two Mind/Body courses, each of which will be held once a week for 8 consecutive weeks. Each class will last 1.5-2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderately severe Ulcerative Colitis
* Age 18-70
* Must have inactive disease at the time of recruitment, with at least one documented disease flare-up within the past 2 years.
* Must be on either no IBD medication or have been on a stable dose of any of the following medications for the specified amount of time: Mesalamine or Sulfasalazine for at least 6 weeks; Remicade for at least 10 weeks; Imuran or Mercaptopurine at stable and unchanged dose for at least 8 weeks.

Exclusion Criteria:

* Active Ulcerative Colitis or daily rectal bleeding for 7 days
* Taking oral steroids within 30 days of enrollment, topical agents (steroids or 5-ASA) within 14 days,immunomodulators such as Methotrexate or Imuran/6-MP and Infliximab within 90 days
* History of colon resection
* Antibiotics use within the previous 14 days
* Pregnant or lactating women
* Significant chronic disorders like severe cardiac disease (NY functional state score>3), renal disease (creatinine>3 mg/dL), pulmonary disease (shortness of breath at rest or need for oxygen use), active infection, or other organ system disease requiring medical visits > 3 times /year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
gut inflammation assessed by stool Calprotectin | (1) initial measurement (2) within 1 month of completion of course (3) 6 months after completion of course (4) 1 year after completion of course

SECONDARY OUTCOMES:
Gut oxidative tissue injury assessed by mucosal protein oxidation (protein carbonyl) | (1) initial measurement (2) within 1 month of completion of course (3) 6 months after completion of course (4) 1 year after completion of course
stress responses assessed by 24h urinary cortisol and psychological questionnaire | (1) initial measurement (2) within 1 month of completion of course (3) 6 months after completion of course (4) 1 year after completion of course
prevention of flare-up assessed by IBD-related clinical, endoscopic, and histological indices | (1) initial measurement (2) within 1 month of completion of course (3) 6 months after completion of course (4) 1 year after completion of course

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keshavarzian, M.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Jedel S, Hoffman A, Merriman P, Swanson B, Voigt R, Rajan KB, Shaikh M, Li H, Keshavarzian A. A randomized controlled trial of mindfulness-based stress reduction to prevent flare-up in patients with inactive ulcerative colitis. Digestion. 2014;89(2):142-55. doi: 10.1159/000356316. Epub 2014 Feb 14. PMID 24557009